CLINICAL TRIAL: NCT01240837
Title: Investigation of the Glycaemic Index of Arenga Pinnata Palm Sugar
Brief Title: Effect of Palm Sugar on Blood Glucose Concentrations
Acronym: LIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 33657
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Adults
Keywords: glycaemic index; arenga pinnata sugar; palm sugar; diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Gur; Glucose; Sucrose; Sugars; Dietary Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- glucose (Active Comparator)
  Interventions: Other: Glucose
- sucrose (Active Comparator)
  Interventions: Other: Sucrose
- palm sugar (Experimental)
  Interventions: Other: Arenga Pinnata Sugar

INTERVENTIONS:
Other: Arenga Pinnata Sugar — 50 g palm sugar given orally 1 time in 250 ml of water. Blood glucose measurements will then be taken at time points, 0, 15, 30, 45, 60, 90 and 120 minutes.
  Other Names: palm sugar
  Arms: palm sugar
Other: Glucose — 50 g glucose given orally 3 time in 250 ml of water. Blood glucose measurements will then be taken at time points, 0, 15, 30, 45, 60, 90 and 120 minutes.
  Arms: glucose
Other: Sucrose — 50 g sucrose given orally 1 time in 250 ml of water. Blood glucose measurements will then be taken at time points, 0, 15, 30, 45, 60, 90 and 120 minutes.
  Other Names: sugar; table sugar
  Arms: sucrose

SUMMARY:
The purpose of this study is to determine by how much, the ingestion of palm sugar increases blood glucose concentrations and what the corresponding glycaemic index is. The investigators estimate that the glycaemic index will be 68 (equal to that of sucrose).

ELIGIBILITY:
Inclusion criteria:

* Healthy: as judged by the participant;
* Age: 18 to 35.

Exclusion criteria:

* Pregnant or lactating females
* Presence of a chronic disease such as diabetes, illness, dysmetabolic syndrome
* 18.5 < BMI < 25
* Allergy or intolerance to palms or coconuts
* Weight loss or gain of more then 5 kg in the last two months
* Fasting blood glucose levels <100 mg/dl or 5.6 mmol/l
* Smokers
* Use of medications other then birth control
* Previous problems with blood sampling

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentrations | 2 months
  During the labratory visits subjects will ingest glucose (control), sucrose or palm sugar. At time points 0, 15, 30, 45, 60, 90 and 120 minutes post ingestion blood glucose concentrations will be measured by finger prick blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Afman, Dr, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands